CLINICAL TRIAL: NCT02232867
Title: Adjunct Locomotor Training to Improve Walking Ability After Stroke
Brief Title: Arm and Leg Cycling Exercise After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Victoria (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Stroke Network (Other)
Responsible Party: Principal Investigator, Dr. E. Paul Zehr, Dr. E. Paul Zehr, University of Victoria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-480-04d
Record Dates: First submitted 2014-08-28; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
Keywords: rehabilitation; stroke; walking; interlimb connections
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm and Leg Cycling Exercise Program (Experimental): Multiple baseline test sessions will be used for the same participant to establish a meaningful baseline thus confirming consistency of all outcome measures prior to the intervention.
  Interventions: Behavioral: Arm and Leg Cycling Exercise Program

INTERVENTIONS:
Behavioral: Arm and Leg Cycling Exercise Program — Participants will perform arm and leg cycling training three times a week, with 30 minutes of aggregate exercise time per session. To evaluate the physiological cost of exercise, heart rate and a rating of perceived exertion will be collected. The progressive element of this training will include increasing the resistance of the ergometer over the six weeks in order to maintain the same relative exercise stress.

SUMMARY:
It has been found that arm and leg cycling is similar to walking in terms of the muscle activation patterns and joint ranges of motion. In addition, arm and leg cycling and walking activate similar neural pathways. Another advantage of arm and leg cycling is that it involves coordination of all four limbs in a rhythmic movement. This may be particularly beneficial given previous findings that arm movement contributes to the activation of leg muscles during walking in humans. This is achieved with interconnected neural pathways that link the arms to the legs. These neural interlimb connections remain intact in stroke victims, such that maximizing the contribution of the arms to the legs may increase coordination for walking. Thus, the objectives of this research are to determine if arm and leg cycling can be used to increase the strength of interlimb connections and if this helps to improve walking ability in a post-stroke population. It is hypothesized that arm and leg cycling will transfer to improvements in walking in a post stroke population.

DETAILED DESCRIPTION:
For those who have suffered a stroke, damage to the brain can result in a decreased ability to walk, thus decreasing quality of life in a significant way. Traditionally, body weight supported treadmill training has been used for walking rehabilitation; however, this therapy requires specialized technicians, equipment, and facilities. Arm and leg cycle ergometers, a device commonly found in a gym, could provide an inexpensive and readily accessible means for walking rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* lives within the Victoria, Vancouver Island, and Vancouver mainland communities

Exclusion Criteria:

* inability to stand for 5 minutes unassisted

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in Treadmill Walking Characteristics | Baseline, immediately post-intervention (average of 4 days following last exercise session)
  Treadmill walking characteristics will be gauged via a customized analysis of muscle activity patterns and lower limb joint kinematics. Walking frequency, symmetry, and timing will also be analyzed

SECONDARY OUTCOMES:
Interlimb Connections | Baseline, immediately post-intervention (average of 4 days following the last exercise session)
  To assess the strength of inter-limb coupling, simultaneous electrical stimulation will be applied to (5x1.0ms trains at 300Hz) the cutaneous nerves in the hand (superficial radial) and foot (superficial peroneal). The reflex responses recorded in all four limbs will be evaluated at different phases of the walking cycle.
Fugl-Meyer Assessment | Baseline, immediately post-intervention (average of 4 days following the last exercise session)
  The Fugl-Meyer Assessment is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Brunnstrom recovery stages | Baseline, immediately post-intervention (average of 4 days following the last exercise session)
  The Brunnstrom Approach emphasises the synergic pattern of movement which develops during recovery from hemiplegia.
Timed up and go test | Baseline, immediately post-intervention (average of 4 days following the last exercise session)
  The Timed Up and Go test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require.
10 meter walk test | Baseline, immediately post-intervention (average of 4 days following the last exercise session)
  The 10 meter walk test is a timed test to evaluate walking speed
Six minute walk test | Baseline, immediately post-intervention (average of 4 days following last exercise session)
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.

CONTACTS AND LOCATIONS:
Overall Officials: E. Paul Zehr, PhD, Principal Investigator — University of Victoria
Locations (1):
- Rehabilitation Neuroscience Laboratory, Victoria, British Columbia, Canada